CLINICAL TRIAL: NCT02260739
Title: Sequential Analysis in Patients With an Hemopathy
Acronym: S-HEMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-A00208-37; 2013/2031 (Other: CSET number)
Record Dates: First submitted 2014-09-16; First posted 2014-10-09 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Hemopathy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- chronic myelomonocytic leukemia (Other): Three cohorts will be investigated: ET (essential thrombocythemia), IMF and secondary MF (myelofibrosis) and CMML (chronic myelomonocytic leukemia)
  Interventions: Other: Blood samples
- essential thrombocytemia (Other): Three cohorts will be investigated: ET (essential thrombocythemia), IMF and secondary MF (myelofibrosis) and CMML (chronic myelomonocytic leukemia)
  Interventions: Other: Blood samples
- myelofibrosis (Other): Three cohorts will be investigated: ET (essential thrombocythemia), IMF and secondary MF (myelofibrosis) and CMML (chronic myelomonocytic leukemia)
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples

SUMMARY:
Recent advances in hematology clearly illustrate that the simple "clonal" nature of various hematological malignancies may not really reflect the reality of malignant cells natural expansion. This has been nicely illustrated in recent works in AML for example where subclones coexists in the same patient at the same time, but could also differentially expand over time because of effects of therapeutics intervention, but also by oncogenic spontaneous events (1).

These observations have been done recently because of next generation sequencing that allows to discriminate in the same tumor samples, different subclones and to analyse the clonal architecture. Sequential analyses could help us to identify the first oncogenic event and to correlate disease progression to the emergence of subclones.

For all these reasons it is of a major interest to precisely understand the architecture of the clone in MPNs, especially to understand which is the initiating event and how from this initial event the clone develops.

In MPNs in which JAK2V617F is the initiating event, its targeting is expected to be extremely effective. If JAK2V617F is a secondary event its targeting might allow to alleviate the MPN, but may favor the development of other malignant hemopathies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a malignant hematological disease.
* Signed written informed consent
* Age and Sex : men and women aged 18 years or older
* Patients affiliated to a social security system

Exclusion Criteria:

- Patients protected by law, in accordance with Articles L1121-L1121-5 to 8 of the Code of Public Health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Identification of new genetic alterations | At baseline and then every 6 months up to 24 months
  Identification of new genetic alterations in patients with hematological malignancies by next generation sequencing using blood samples

SECONDARY OUTCOMES:
Sequential analysis of the malignant clones | At baseline and 12 months after inclusion
  Sequential analysis of the malignant clones for each patient included in the trial using genetic markers

CONTACTS AND LOCATIONS:
Overall Officials: Vincent RIBRAG, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France